CLINICAL TRIAL: NCT06510452
Title: Efficacy of Antibiotic Prophylaxis in Metabolic Bariatric Surgery: A Randomized Controlled Trial
Brief Title: Antibiotic Prophylaxis in Metabolic Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, head of bariatric surgery, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AB-BAR-2024
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Antibiotic Reaction; Wound Infection Superficial; Wound Infection Deep; Bariatric Surgery Candidate; Complication,Postoperative
Keywords: anti-biotics; non-inferiority; surgical side infection
MeSH Terms: conditions — Postoperative Complications | interventions — Cefazolin; Metronidazole; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NACL0.9% (Experimental): Group A will receive 100 ml NACL0.9% without any antibiotics in it.
  Interventions: Drug: NACL 0.9% 100 ml
- Cefazolin +Metronidazole (Active Comparator): Group B will receive 2000 mg of Cefazolin and 500 mg of Metronidazole IV dissolved in 100 ml NACL0.9%. Both antibiotics will be administered at least 30 minutes before surgery to ensure adequate tissue concentrations at the time of incision.
  Interventions: Drug: 2000 mg of Cefazolin; Drug: 500 mg of Metronidazole IV

INTERVENTIONS:
Drug: 2000 mg of Cefazolin — receive 2000 mg of Cefazolin and 500 mg of Metronidazole IV dissolved in 100 ml NACL0.9%.
  Other Names: Kefzol
  Arms: Cefazolin +Metronidazole
Drug: 500 mg of Metronidazole IV — receive 2000 mg of Cefazolin and 500 mg of Metronidazole IV dissolved in 100 ml NACL0.9%.
  Other Names: Flagyl
  Arms: Cefazolin +Metronidazole
Drug: NACL 0.9% 100 ml — receive 100 ml NACL0.9% without any antibiotics in it.
  Other Names: Saline
  Arms: NACL0.9%

SUMMARY:
SUMMARY Rationale: Prophylactic antibiotics in laparoscopic surgeries, including Metabolic Bariatric Surgery (MBS), are routinely provided to reduce postoperative infections, especially at wound incision sites. However, since incisional wound infections in laparoscopic MBS are rare and morbidity is very low, the benefit of antibiotic prophylaxis is questionable.

Objective: Evaluate the non-inferiority of omitting antibiotic prophylaxis in MBS. Compare postoperative outcomes between Group A (no antibiotics) and Group B (standard antibiotic care) to determine if omission increases complications, particularly wound infections.

Study Design: Randomized controlled trial (RCT), double-blind.

Study Population: Patients with obesity eligible for MBS.

Intervention:

* Group A (No Antibiotic Prophylaxis): Undergo MBS without antibiotics to test safety regarding postoperative complications, focusing on surgical site infections (SSIs).
* Group B (Standard Antibiotic Prophylaxis): Receive standard one-time antibiotics before incision.

Main Study Parameters/Endpoints: Compare the incidence of incisional and organ/space SSIs within six weeks post-surgery between Group A and Group B to determine if omitting antibiotics affects infection rates.

DETAILED DESCRIPTION:
Nature and Extent of the Burden and Risks:

Rationale:

1. Cost-Effectiveness: Reducing antibiotic use could lower surgical costs.
2. Resource Utilization: Simplifying protocols save hospital resources.
3. Antibiotic Resistance: Reducing use helps combat resistant bacteria.
4. Adverse Reactions: Fewer antibiotics may reduce side effects.

Risk Assessment:

1. Increased Infection Rates: Monitor SSI and organ/space SSI rates closely.
2. Anastomotic Leaks and Reoperations: Assess the impact on leaks and operations.
3. Readmissions and Postoperative Interventions: Evaluate the effect on readmission and intervention rates.

Group Relatedness:

Comparing groups with and without antibiotics provides evi-dence-based insights into the safety of modifying standard practices to optimize health outcomes and resource use.

ELIGIBILITY:
Inclusion Criteria:

° Patients must be older than 18 and meet the eligibility criteria for MBS as outlined by the International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) and the Dutch Federation of Medical Specialists for the surgical treatment of obesity.

Exclusion Criteria:

* Patients undergoing immunotherapy or corticosteroid treatment for Crohn's disease or rheumatoid arthritis.
* Patients with a history of endocarditis require prophylactic antibiotics.
* Patients with known severe allergies to antibiotics.
* Patients with active infections or recently treated with antibiotics (within the last 30 days).
* Patients with compromised immune systems, including those with HIV/AIDS or undergoing chemotherapy.
* Patients with chronic liver or kidney disease.
* Patients with uncontrolled diabetes (HbA1c > 9%).
* Patients with a history of previous metabolic bariatric surgery.
* Pregnant or breastfeeding women.
* Patients with any other medical condition that, in the opinion of the investigator, would compromise the patient's safety or the study's integrity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3352 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of incidence of postoperative wound infections in both treatment arms | until 6 weeks post operative
  Aims to evaluate the non-inferiority of foregoing antibiotic prophylaxis in MBS. The study will compare postoperative outcomes between two groups: Group A, which will not receive antibiotic prophylaxis, and Group B, which will receive standard care including a one-time administration of antibiotics, to test the hypothesis that omitting antibiotic prophylaxis does not significantly increase the incidence of postoperative complications, in particular wound infections.

CONTACTS AND LOCATIONS:
Locations (2):
- Madina Women's Hospital, Alexandria, Egypt
- WeightWorks clinics, Amersfoort, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after the completion of the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com) and handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers, where all the research data were stored, are certified according to ISO27001, ISO9001, and Dutch NEN7510.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the study been peer-reviewed for 20 years available.
Access Criteria: contact the corresponding author

REFERENCES:
- [Background] CDC antimicrobial resistance. Available from: https://www.cdc.gov/drugresistance/about.html
- [Result] Aktas A, Kayaalp C, Gunes O, Kirkil C, Tardu A, Aydin MC, Bag YM, Cayci HM, Arslan U, Sumer F, Aygen E. Surgical Site Infections after Laparoscopic Bariatric Surgery: Is Routine Antibiotic Prophylaxis Required? Surg Infect (Larchmt). 2021 Sep;22(7):705-712. doi: 10.1089/sur.2020.426. Epub 2021 Jan 8. PMID 33416442
- [Result] Dang JT, Tran C, Switzer N, Delisle M, Laffin M, Madsen K, Birch DW, Karmali S. Predicting surgical site infections following laparoscopic bariatric surgery: development of the BariWound tool using the MBSAQIP database. Surg Endosc. 2020 Apr;34(4):1802-1811. doi: 10.1007/s00464-019-06932-6. Epub 2019 Jun 24. PMID 31236724
- [Result] Shope TR, Cooney RN, McLeod J, Miller CA, Haluck RS. Early results after laparoscopic gastric bypass: EEA vs GIA stapled gastrojejunal anastomosis. Obes Surg. 2003 Jun;13(3):355-9. doi: 10.1381/096089203765887651. PMID 12841893
- [Result] Alasfar F, Sabnis A, Liu R, Chand B. Reduction of circular stapler-related wound infection in patients undergoing laparoscopic Roux-en-Y gastric bypass, Cleveland clinic technique. Obes Surg. 2010 Feb;20(2):168-72. doi: 10.1007/s11695-008-9708-3. Epub 2008 Oct 7. PMID 18839083
- [Result] Schauer PR, Ikramuddin S, Gourash W, Ramanathan R, Luketich J. Outcomes after laparoscopic Roux-en-Y gastric bypass for morbid obesity. Ann Surg. 2000 Oct;232(4):515-29. doi: 10.1097/00000658-200010000-00007. PMID 10998650
- [Result] Finks JF, Carlin A, Share D, O'Reilly A, Fan Z, Birkmeyer J, Birkmeyer N; Michigan Bariatric Surgery Collaborative from the Michigan Surgical Collaborative for Outcomes Research Evaluation. Effect of surgical techniques on clinical outcomes after laparoscopic gastric bypass--results from the Michigan Bariatric Surgery Collaborative. Surg Obes Relat Dis. 2011 May-Jun;7(3):284-9. doi: 10.1016/j.soard.2010.10.004. Epub 2010 Oct 16. PMID 21126927
- [Result] Mangram AJ, Horan TC, Pearson ML, Silver LC. Guideline for Prevention of Surgical Site Infection, 1999. 1999;27.
- [Result] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists (ASHP); Infectious Diseases Society of America (IDSA); Surgical Infection Society (SIS); Society for Healthcare Epidemiology of America (SHEA). Clinical practice guidelines for antimicrobial prophylaxis in surgery. Surg Infect (Larchmt). 2013 Feb;14(1):73-156. doi: 10.1089/sur.2013.9999. Epub 2013 Mar 5. No abstract available. PMID 23461695
- [Result] Anderson DJ, Podgorny K, Berrios-Torres SI, Bratzler DW, Dellinger EP, Greene L, Nyquist AC, Saiman L, Yokoe DS, Maragakis LL, Kaye KS. Strategies to prevent surgical site infections in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Sep;35 Suppl 2:S66-88. doi: 10.1017/s0899823x00193869. No abstract available. PMID 25376070
- [Result] De Luca M, Angrisani L, Himpens J, Busetto L, Scopinaro N, Weiner R, Sartori A, Stier C, Lakdawala M, Bhasker AG, Buchwald H, Dixon J, Chiappetta S, Kolberg HC, Fruhbeck G, Sarwer DB, Suter M, Soricelli E, Bluher M, Vilallonga R, Sharma A, Shikora S. Indications for Surgery for Obesity and Weight-Related Diseases: Position Statements from the International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO). Obes Surg. 2016 Aug;26(8):1659-96. doi: 10.1007/s11695-016-2271-4. No abstract available. PMID 27412673
- [Result] Eisenberg D, Shikora SA, Aarts E, Aminian A, Angrisani L, Cohen RV, de Luca M, Faria SL, Goodpaster KPS, Haddad A, Himpens JM, Kow L, Kurian M, Loi K, Mahawar K, Nimeri A, O'Kane M, Papasavas PK, Ponce J, Pratt JSA, Rogers AM, Steele KE, Suter M, Kothari SN. 2022 American Society of Metabolic and Bariatric Surgery (ASMBS) and International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) Indications for Metabolic and Bariatric Surgery. Obes Surg. 2023 Jan;33(1):3-14. doi: 10.1007/s11695-022-06332-1. PMID 36336720
- [Result] Joint Task Force on Practice Parameters; American Academy of Allergy, Asthma and Immunology; American College of Allergy, Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. Drug allergy: an updated practice parameter. Ann Allergy Asthma Immunol. 2010 Oct;105(4):259-273. doi: 10.1016/j.anai.2010.08.002. PMID 20934625
- [Result] Jourdan A, Sangha B, Kim E, Nawaz S, Malik V, Vij R, Sekhsaria S. Antibiotic hypersensitivity and adverse reactions: management and implications in clinical practice. Allergy Asthma Clin Immunol. 2020 Jan 21;16:6. doi: 10.1186/s13223-020-0402-x. eCollection 2020. PMID 31993070
- [Result] WHO antimicrobial resistance. Available from: https://www.who.int/news-room/fact-sheets/detail/antimicrobial-resistance
- [Result] Mokrani D, Chommeloux J, Pineton de Chambrun M, Hekimian G, Luyt CE. Antibiotic stewardship in the ICU: time to shift into overdrive. Ann Intensive Care. 2023 May 6;13(1):39. doi: 10.1186/s13613-023-01134-9. PMID 37148398